CLINICAL TRIAL: NCT04232904
Title: Effect of Transversus Abdominis Plane Block With Bupivacaine on Anti-inflammatory Response in Living Liver Donors
Brief Title: Effect of Transversus Abdominis Plane Block on Anti-inflammatory Response
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Mehmet Ali Erdoğan, Clinical Professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: MAE7
Record Dates: First submitted 2019-12-17; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Liver Transplant; Complications; Inflammatory Response
Keywords: living liver donor; TAP block; cytokine; bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP Block Group (Active Comparator): this is study group.
  Interventions: Procedure: Transversus abdominous plane block (TAP Block)
- Control Group (No Intervention): This patients are control group. TAP block will be not perform

INTERVENTIONS:
Procedure: Transversus abdominous plane block (TAP Block) — TAP block which is a peripheral nerve block preferred to postoperative pain management.
  Arms: TAP Block Group

SUMMARY:
The liver transplantation is the only treatment for end-stage liver failure. Lack of sufficient organs from the cadaver to meet the organ needs has increased the interest in a live organ donor transplantation. A peripheral nerve block, transversus abdominous plane block (TAP block); When combined with general anesthesia in live liver donors, it has been shown to significantly reduce perioperative and postoperative opioid consumption, provide shorter recovery time and shorten hospital stay. It has been shown that regional block techniques using local anesthetics and analgesic adjuvants modulate both local and systemic inflammatory reactions caused by surgical injury. Cytokines are important mediators of local and systemic inflammatory response including hyperalgesia after surgery. In literature, the effect of TAP block on anti-inflammatory cytokines in live liver donors was not shown. The aim of this study is to investigate the effect of bupivacaine TAP block on antiflammatory response in living liver donors.

DETAILED DESCRIPTION:
The liver transplantation is the only treatment for end-stage liver failure. Lack of sufficient organs from the cadaver to meet the organ needs has increased the interest in a live organ donor transplantation. A peripheral nerve block, transversus abdominous plane block (TAP block); When combined with general anesthesia in live liver donors, it has been shown to significantly reduce perioperative and postoperative opioid consumption, provide shorter recovery time and shorten hospital stay.Immunological, metabolic and endocrine reactions occur due to tissue damage, pain and anesthesia caused by surgery. It has been shown that regional block techniques using local anesthetics and analgesic adjuvants modulate both local and systemic inflammatory reactions caused by surgical injury. Cytokines are important mediators of local and systemic inflammatory response including hyperalgesia after surgery. Cytokines are indispensable for wound healing and restoration of homeostasis, but usually the overactivity of either proinflammatory or anti-inflammatory cytokines damages the host. With Preemptive epidural analgesia, peripheral nerve block and thoracic epidural analgesia; postoperative pain and proinflammatory cytokines have been reduced. In literature, the effect of TAP block on anti-inflammatory cytokines in live liver donors was not shown. The aim of this study is to investigate the effect of bupivakine TAP block on antiinflammatory response in live liver donors.This prospective clinical study will performs in 72 liver transplant donors aged 18-65 years, ASA I-II, schedule for right hepatectomy surgery. Peripheral vascular access will open and blood samples will take for preoperative cytokine and bupivacaine measurements.The primary aim of this study was to investigate the effect of TAP block on the inflammatory response by cytokine level. The secondary aim of this study is to determine the plasma bupivacaine concentrations in patients undergoing TAP block and to investigate the relationship between plasma bupivacaine level and cytokine levels.

ELIGIBILITY:
Inclusion Criteria:

* liver transplant donors schedule for right hepatectomy surgery.
* aged 18-65 years,

Exclusion Criteria:

* systemic disease (such as diabetes and hypertension),
* used opioid or NSAID in the last week,
* coagulation pathology,
* a history of allergy to drugs used in the study
* refusal to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is not based on self-representation of gender identity.
Enrollment: 70 (Estimated)
Dates: Start 2019-12-02 (Actual); Primary Completion 2020-06-15 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
cytokine level (interleukine-1, interleukine-6, tumor necrosis factor) | Change from baseline cytokines levels at 24 hours postoperatively
  Immunological, metabolic and endocrine reactions occur due to tissue damage, pain and anesthesia caused by surgery. Cytokines are important mediators of local and systemic inflammatory response including hyperalgesia after surgery. Cytokines are indispensable for wound healing and restoration of homeostasis, but usually the overactivity of either proinflammatory or anti-inflammatory cytokines damages the host.

SECONDARY OUTCOMES:
correlation of plasma bupivacaine level and cytokine level | Change from baseline correlation of plasma bupivacaine level and cytokines levels at 24 hours postoperatively
  The relationship between plasma bupivacaine level and cytokine level in patients undergoing TAP block
The plasma bupivacaine concentrations | Change from baseline plasma bupivacaine concentrations at 24 hours postoperatively
  The plasma bupivacaine concentrations in patients undergoing TAP block

CONTACTS AND LOCATIONS:
Overall Officials: Ulku Ozgul, MD, Principal Investigator — Inonu University, Scholl of Madicine, Malatya Turkey
Locations (1):
- Inonu university, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bagry H, de la Cuadra Fontaine JC, Asenjo JF, Bracco D, Carli F. Effect of a continuous peripheral nerve block on the inflammatory response in knee arthroplasty. Reg Anesth Pain Med. 2008 Jan-Feb;33(1):17-23. doi: 10.1016/j.rapm.2007.06.398. PMID 18155052
- [Result] Kitlik A, Erdogan MA, Ozgul U, Aydogan MS, Ucar M, Toprak HI, Colak C, Durmus M. Ultrasound-guided transversus abdominis plane block for postoperative analgesia in living liver donors: A prospective, randomized, double-blinded clinical trial. J Clin Anesth. 2017 Feb;37:103-107. doi: 10.1016/j.jclinane.2016.12.018. Epub 2017 Jan 7. PMID 28235493